CLINICAL TRIAL: NCT04941196
Title: A Single Centre, Cross-over, Single Dose, Two Period, Randomized, Open Label Bioequivalence Study of Anplag® 90mg (Ticagrelor) Tablet With Brilinta® 90 mg (Ticagrelor) Tablet in Healthy Adult Male Pakistani Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Anplag® 90mg (Ticagrelor) Tablet & Brilinta® 90 mg (Ticagrelor) Tablet in Healthy Adult Male Pakistani Subjects Under Fasting Condition
Acronym: BE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: PharmEvo Private Limited., Pakistan (Unknown)
Responsible Party: Principal Investigator, Dr. Muhammad Raza Shah, Professor, University of Karachi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CB-030-TIC-2019/Protocol/2.0
Record Dates: First submitted 2021-06-19; First posted 2021-06-28 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Healthy Individuals
Keywords: Bioequivalence Study; Pakistani Population; Bioavailability comparison
MeSH Terms: interventions — Ticagrelor

STUDY DESIGN:
Intervention Model Description: single centre, cross over, single dose, two period, randomized, open label Bioequivalence Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Oral administration of Anplag® 90mg (Ticagrelor) whole Tablet, manufactured by PharmEvo Private Laboratories (Pak) Ltd., after at least 10 hours fast together with 240 mL of ambient temperature water at their scheduled dosing time-point.
  Interventions: Drug: Anplag (Ticagrelor 90 mg)
- Reference Group (Active Comparator): Oral administration of Brilinta® 90mg (Ticagrelor) Whole Tablet, manufactured by AstraZeneca Pharmaceuticals., after at least 10 hours fast together with 240 mL of ambient temperature water at their scheduled dosing time-point.
  Interventions: Drug: Brilinta (Ticagrelor 90 mg)

INTERVENTIONS:
Drug: Anplag (Ticagrelor 90 mg) — Ticagrelor 90 mg Immediate Release tablet
  Arms: Test Group
Drug: Brilinta (Ticagrelor 90 mg) — Ticagrelor 90 mg Immediate Release tablet
  Arms: Reference Group

SUMMARY:
Single oral administration of study drugs (i.e. Anplag® & Brilinta®) in Two periods after at least 10 hours fasting. The periods will be separated by a washout period of 7 days. The purpose of this study is to compare the bioavailability of Anplag® 90mg (Ticagrelor) Tablet with Brilinta® 90 mg (Ticagrelor) Tablet under fasting conditions in healthy Pakistani male subjects.

DETAILED DESCRIPTION:
The subjects will be randomly assigned in period 1 to T or R sequence and will be administered the study drugs T (Anplag® 90 mg) or R (Brilinta® 90 mg) with 240 mL ambient temperature water following at least 10 hours fasting. Blood samples will be withdrawn at pre-determined time points for estimation of plasma drug concentration upto 48 hours post dose. the subjects will be crossed over in Period 2 separated by a washout period of 7 days and administered RT sequence in period 2. Similar procedure of blood sampling will be applied for estimation of plasma drug concentration upto 48 hours post dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged 18 to 55 years inclusive.
* Subjects with a body mass index from 18.5 to 30.0 kg/m2.
* Subjects who are healthy as determined by routine physical examination, including vital sign monitoring (i.e., blood pressure, heart rate, and temperature), 12-lead ECG and laboratory analysis (i.e., hematology, blood biochemistry, Serology and urinalysis), or as determined by the investigator.
* Subjects should have negative urine test for drugs of abuse (Opiates and cannabinoids will be tested) and negative result for alcohol breath test at screening and prior to each check-in
* Tested negative for COVID-19 (through COVID-19 antibody testing).
* Subjects and their partners are willing to use reliable non-hormonal contraceptive methods (condoms, diaphragm, non-hormonal intra-uterine device (IUD), female or male sterilization or sexual abstinence) throughout the study and up to 30 days after the last administration of the study drug.
* All subjects should be free from any epidemic or contagious disease (e.g. Malaria, Dengue, COVID-19).
* Subjects are able to, understand and sign the Informed Consent Form for Medical Screening during their screening visit and Participation Informed Consent Form on study Check-In day
* Subject agreed not to consume food or beverages like tea, coffee, cola drinks, chocolates containing Xanthene derivatives (including caffeine, theobromines, etc.) and/or poppy seeds (Khashkhash) within 48-hours prior to drug administration until last blood draw in each study period.
* Subject agreed not to intake prescription medicine within 14 days or 5 half-lives (whichever is longer) prior to first dose of study medicine.
* Subject agreed not to intake non-prescription drugs (OTC such as aspirin, ibuprofen, naproxen, non-steroidal anti-inflammatory drugs (NSAIDs), or any other drug known to increase the tendency for bleeding within 14 days prior to first dose of study medicine.
* Subject agreed to discontinue vitamins, dietary and herbal supplements within 14 days prior to the first dose of study medication.
* Subject agreed not to consume grapefruit and/or its products within 14 days prior to the start of study.

Exclusion Criteria:

* Refused to sign Informed Consent Form.
* Inability to take oral medication.
* Tested positive for COVID-19 (through COVID-19 antibody testing).
* History of smoking (> 5 cigarette/day), alcoholism, and positive test for drug of abuse.
* Heavy pan or gutka user as judged by teeth/mouth inspection.
* Subjects with clinically relevant evidence of cardiovascular, gastrointestinal/hepatic, renal, psychiatric, respiratory, urogenital, hematologic/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, drug hypersensitivity, allergy, endocrine, major surgery or other relevant diseases as revealed by medical history, physical examination, and laboratory assessments which may interfere with the absorption, distribution, metabolism or elimination of drugs or constitute a risk factor when taking study medication.
* Donation or loss of more than 450 mL of blood within 3 months prior to the screening.
* History of intake of any prescribed medicine during a period of 30 days, prior to drug administration day of study.
* Subject is allergic to Ticagrelor and/or other antiplatelet medications/platelet aggregation inhibitors.
* Subject has received any investigational drug within four weeks prior to screening.
* Subjects whose heart rate is abnormally low (usually lower than 60 beats per minute) and subject already have in place a device that paces the heart (pacemaker).
* Subjects with a history of hemophilia, von Willebrand's disease, lupus anticoagulant, or other diseases/syndromes that can either alter or increase the propensity for bleeding.
* A personal history of vascular abnormalities including aneurysms; a personal history of severe hemorrhage, non-traumatic bleeding, bleeding risks, hematemesis, melena, hemoptysis, severe epistaxis, severe thrombocytopenia, intracranial hemorrhage; or rectal bleeding within 1 year prior to screening; or history suggestive of peptic ulcer disease; or at the discretion of the investigator.
* Platelet count is less than 150 x 10^9/L.
* Subject has had a blood test that showed more than the usual amount of uric acid.
* Subjects receiving oral anticoagulants often referred to as "blood thinners" which include warfarin.
* History of any significant illness in the last four weeks .
* Consumption of grapefruit and/or its products within 14 days prior to the start of study.
* Subjects who test positive for syphilis (VDRL) or who are known to have serum hepatitis or who are carriers of the Hepatitis B surface antigen (HBs Ag) or are carriers of antibodies to hepatitis C virus (anti-HCV), human immunodeficiency virus (HIV-1 or HIV-2) or COVID-19.
* Individuals having undergone any major surgery (including dental work) within 3 months prior to the start of the study, unless deemed eligible, otherwise by the Principal Investigator or whomever he/she may designate.
* Subject has a history of any illness that, in the opinion of investigator might confound the result of the study or pose any risk in administrating Ticagrelor to the subject.
* Subjects with any condition, which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or elimination of drugs.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy adult Pakistani Male subjects
Enrollment: 30 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-48 hours post dose
  Maximum Plasma Drug concentration
Tmax | 0-48 hours post dose
  Time required to reach maximum plasma Ticagrelor concentration
AUC | 0-48 hours post dose
  Area under the plsama drug concentration versus time curve

SECONDARY OUTCOMES:
Blood pressure | 0-48 hours post dose
  monitoring of blood pressure at specified time intervals
Heart rate | 0-48 hours post dose
  Monitoring of Heart rate at pre-specified time intervals
Body temprature | 0-48 hours post dose
  measurement of body temperature at pre-determined time intervals

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Muhammad R Shah, PhD, Principal Investigator — Center for bio-equivalence studies and clinical research, ICCBS, University of Karachi, Pakistan; Dr. Naghma Hashmi (Co-PI), PhD, Principal Investigator — Center for bio-equivalence studies and clinical research, ICCBS, University of Karachi, Pakistan
Locations (1):
- Center for Bioequivalence Studies and clinical research, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be obtained upon proper request to principal investigator unless the volunteer's confidentiality is not compromised.

REFERENCES:
- [Derived] Hashmi N, Jawaid M, Shah MR. Bioequivalence assessment of two Ticagrelor formulations under fasting condition in healthy Pakistani subjects. Pak J Med Sci. 2023 Nov-Dec;39(6):1647-1651. doi: 10.12669/pjms.39.6.8203. PMID 37936786